CLINICAL TRIAL: NCT06789107
Title: Clinical Trial of Blinatumomab in Refractory/Active Systemic Lupus Erythematosus in Children
Brief Title: Blinatumomab in Refractory Active Childhood Systemic Lupus Erythematosus
Acronym: BRASLE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mao Jianhua (Other)
Responsible Party: Sponsor-Investigator, Mao Jianhua, Professor, The Children's Hospital of Zhejiang University School of Medicine
Organization: The Children's Hospital of Zhejiang University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRASLE
Record Dates: First submitted 2024-12-05; First posted 2025-01-23 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus (SLE); Children; Blinatumomab
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: Blinatumomab Treatment (Experimental): Blinatumomab treatment for Refractory/Active Systemic Lupus Erythematosus. Patients will receive two 5-day cycles of Blinatumomab (5 µg/m²/day, maximum dose 9 µg/day), administered intravenously. The second cycle will begin on the first day of the third week following the first cycle.
  Interventions: Drug: Blinatumomab 9ug

INTERVENTIONS:
Drug: Blinatumomab 9ug — Blinatumomab for Refractory/Active Systemic Lupus Erythematosus. Patients will receive two 5-day cycles of Blinatumomab (5 µg/m²/day, maximum dose 9 µg/day), administered intravenously. The second cycle will begin on the first day of the third week following the first cycle.

SUMMARY:
The goal of this clinical trial is to learn if blinatumomab works to treat refractory or active systemic lupus erythematosus (SLE) in children and adults. It will also learn about the safety of blinatumomab. The main questions it aims to answer are:

Does blinatumomab improve symptoms and disease activity in refractory/active SLE? What side effects or adverse events do participants experience when taking blinatumomab?

Participants will:

Receive two courses of blinatumomab injections over five consecutive days each Be monitored for 52 weeks to evaluate the treatment's safety and effectiveness Undergo regular blood tests and assessments of disease activity during follow-up visits Researchers will collect data on changes in serological markers, disease symptoms, and adverse events throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be eligible for enrollment:

1. Age: ≥ 5 years old.
2. Diagnosis: Diagnosed with systemic lupus erythematosus (SLE) based on the 2019 EULAR/ACR classification criteria.
3. Positive Antibody: At least one of the following antibodies positive within 12 months before screening or during the screening period:

   * Antinuclear antibody (ANA) ≥ 1:80.
   * Anti-double-stranded DNA (anti-dsDNA) antibody above the upper limit of normal (ULN).
   * Anti-Smith (Anti-Sm) antibody above the ULN.
4. Treatment Resistance: Inadequate response to at least three of the following:

   * Oral corticosteroids (OCS),
   * Antimalarials,
   * Conventional immunosuppressants (e.g., cyclophosphamide, mycophenolate mofetil, azathioprine, methotrexate, cyclosporine, tacrolimus, sirolimus, leflunomide),
   * Biologics (e.g., TULIP-2, belimumab, rituximab). At least one treatment must involve immunosuppressants or biologics.
5. SLEDAI-2000 Score: ≥ 6 based on the SLEDAI-2000 scoring system.
6. Stable Standard Treatment: Currently receiving one or more of the following treatments at a stable dose:

   * OCS (e.g., prednisone acetate or equivalent) at a stable dose for ≥7 days prior to initiation;
   * Antimalarials: Dose stable for at least 7 days prior to the first dose.
   * Conventional immunosuppressants: Stable dose for at least 4 weeks before screening and throughout the study.
7. Laboratory Parameters:

   * Absolute lymphocyte count (ALC) ≥ 0.5 × 10⁹/L.
   * Peripheral CD19+ B cell count ≥ 25 cells/μL.
   * Absolute neutrophil count (ANC) ≥ 0.5 × 10⁹/L.
   * Hemoglobin ≥ 80 g/L.
   * Platelet count ≥ 75 × 10⁹/L *.
   * Left ventricular ejection fraction (LVEF) ≥ 55% with no significant ECG abnormalities.
   * Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73m².
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN; total bilirubin ≤ 2 × ULN.
   * No severe pulmonary lesions, SpO₂ ≥ 92%.
8. Contraception: Female participants of childbearing potential must have a negative urine pregnancy test and agree to use effective contraception during the study and for 1 year after infusion.
9. Informed Consent: The participant and their legal guardian must provide written informed consent, demonstrating understanding of the study objectives and willingness.

   * Note: For SLE patients with thrombocytopenia below the inclusion threshold due to immune-related causes, and without active bleeding, investigators may use clinical discretion to determine eligibility.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded:

1. Central nervous system disease: active or unstable lupus-related neuropsychiatric disease within 60 days, including epilepsy, confusion, cerebrovascular events, etc.;
2. Acute severe nephritis: renal replacement therapy within 3 months before the screening period or ongoing, or significant kidney disease that, in the opinion of the investigator, may occur and lead to the need for high-dose glucocorticoid (prednisone dose ≥ 2 mg/kg/d or equivalent of other hormones), cyclophosphamide or escalated MMF treatment within the first 3 months of the study;
3. Severe antiphospholipid syndrome within 12 months before or during screening；
4. Congenital heart disease or a history of acute myocardial infarction within 6 months before screening, or severe arrhythmia (including polymorphic ventricular tachycardia, ventricular tachycardia, etc.); or combined with moderate to large pericardial effusion, severe myocarditis, etc.; or unstable vital signs, patients who need blood pressure-raising drugs to maintain blood pressure;
5. Suffering from other diseases that require long-term administration of glucocorticoids or immunosuppressive agents;
6. Having active infections or uncontrollable infections that require systemic treatment within one week before screening;
7. Having received solid organ transplantation or hematopoietic stem cell transplantation within three months before screening; or having grade 2 or higher acute graft-versus-host disease (GVHD) within two weeks before screening;
8. History of severe recurrent or chronic infections, especially recurrent or chronic infections associated with respiratory problems.
9. Immunoglobulin G levels below the lower limit (5-8 years: <4.5 g/L, 9 years and older: <6.0 g/L);
10. History of hepatitis B virus (HBV) infection or positive serology indicating current or past HBV infection. Human immunodeficiency virus (HIV; positive HIV antibody test) and active hepatitis C virus (HCV) infection (detectable HCV ribonucleic acid [RNA]). Active cytomegalovirus (CMV) or Epstein-Barr virus (EBV) infection;
11. A history of tuberculosis or active tuberculosis; or latent tuberculosis treated before the baseline; or subjects with an indeterminate test result who screened positive for PPD or T-spot can be retested, but if the repeat test is also indeterminate, they are excluded;
12. Had a history of macrophage activation syndrome within 1 month prior to screening;
13. Had received any anti-CD19 or anti-CD20 therapy, such as rituximab, obinutuzumab, ocrelizumab, or ofatumumab, within 3 months prior to screening or during screening;
14. Received a JAK inhibitor, Bruton tyrosine kinase (BTK) inhibitor, or tyrosine kinase 2 (TYK2) inhibitor, such as baricitinib, tofacitinib, upadacitinib, filgotinib, ibrutinib, or zanubrutinib and Fenebrutinib, during screening;
15. Treatment with cyclophosphamide or a biologic agent within 4 weeks prior to enrollment, including but not limited to adalimumab, etanercept, golimumab, infliximab, Infliximab), Belimumab, Ustekinumab, Anifrolumab, Secukinumab, or Atacicept;
16. Intolerance or contraindication to the investigational therapy, including a history of severe allergies or allergic reactions to monoclonal antibodies, or a known hypersensitivity to any of the ingredients in belimumab injection;
17. Live vaccine within 4 weeks prior to screening;
18. Positive blood pregnancy test;
19. Patients with known malignant diseases such as tumors before screening;
20. Patients who have participated in other clinical trials within 3 months prior to enrollment;
21. Patients with depression or suicidal tendencies;
22. Other situations where the investigator believes the patient is not suitable for participation in the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-12-08 (Actual); Primary Completion 2027-12-07 (Estimated); Study Completion 2027-12-07 (Estimated)

PRIMARY OUTCOMES:
safety of Blinatumomab | with 12 weeks of Blinatumomab treatment
  Safety and tolerability: type, frequency and severity of adverse events

SECONDARY OUTCOMES:
Proportion of patients achieving DORIS remission after treatment of Blinatumomab | with 24 weeks of Blinatumomab
  DORIS response rate
Proportion of patients achieving SRI-4 remission after treatment of Blinatumomab | 12 weeks and 24 weeks
  SRI-4 response rate
Changes in peripheral blood CD19+ B cells | within 52 weeks
  B cell clearance at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Mao, PhD, MD, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China